CLINICAL TRIAL: NCT07127744
Title: Determination of the Relationship Between Orthodontic Malocclusion Severity and Periodontitis Risk Using RANKL, OPG and Oxidative Stress Markers
Brief Title: Relationship Between Malocclusion Severity and Periodontitis Risk
Status: Not yet recruiting | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek KARADOĞAN, Assoc. Prof. Dr., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: periortho05/2025
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Malocclusion
Keywords: malocclusion; periodontitis; RANKL; Osteoprotegerin; oxidative stress
MeSH Terms: conditions — Malocclusion; Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Gingival Crevicular Fluid (GCF) Collection After isolating the teeth with a cotton roll, supragingival plaque will be removed and a gentle airflow will be used to dry the teeth. GCF samples will be collected by inserting PerioPaper strips into the mesiobuccal gingival sulcus to a depth of approximately 1 mm for 30 seconds. A calibrated Periotron 8000 instrument will then be used to measure the total GCF volume. PerioPaper strips will then be stored at -80°C for future measurements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with normal or minor malocclusion: Patients with a Dental Aesthetic Index Score of ≤25
- Moderate malocclusion: Patients with a Dental Aesthetic Index Score of 26-30
- Severe malocclusion: Patients with a Dental Aesthetic Index Score of 31-35
- Obstructive malocclusion: Patients with a Dental Aesthetic Index Score ≥ 36

SUMMARY:
The goal of this observational study is to examine the potential relationship between the severity of orthodontic malocclusion and the risk of developing periodontitis in individuals by evaluating salivary and gingival crevicular levels of RANKL, osteoprotegerin (OPG), and oxidative stress biomarkers.

The main question it aims to answer is:

Does increasing severity of orthodontic malocclusion contribute to a higher risk of periodontitis through changes in RANKL/OPG balance and oxidative stress levels?

Participants with different levels of tooth misalignment (malocclusion) will be examined to assess the condition of their teeth and gums. During this examination, information such as dental plaque, gum bleeding, and the depth of gum pockets will be recorded. In addition, fluid samples collected from the gums will be tested in the laboratory to measure certain biological substances and chemical markers related to the body's balance between harmful and protective effects. These measurements will be done using special laboratory tests.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the potential relationship between the severity of orthodontic malocclusion and the risk of developing periodontitis through the analysis of RANKL, osteoprotegerin (OPG), and oxidative stress biomarkers. The mechanical effects of malocclusion on teeth and surrounding tissues may lead to inflammation and tissue destruction within the periodontal structures. Understanding the biomolecular mechanisms involved in this process is essential for early diagnosis and preventive approaches.

This cross-sectional study will include individuals with varying degrees of malocclusion severity. Orthodontic status will be determined through clinical evaluation and standardized indices, while periodontal status will be assessed using parameters such as the plaque index, papillary bleeding index, and probing pocket depth. In addition, gingival crevicular fluid (GCF) samples will be collected from participants to measure levels of RANKL, OPG, total antioxidant capacity (TAC), and total oxidative status (TOS) using the ELISA method.

The data obtained will help reveal whether orthodontic abnormalities increase the risk of periodontal disease and how this risk correlates with biomarker levels. The study emphasizes the importance of a holistic evaluation of both orthodontic and periodontal health.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 12 and 18,
* Patients with all permanent teeth,
* Not having taken antibiotics, steroids, and/or nonsteroidal anti-inflammatory drugs in the last 3 weeks,
* Not having an active infectious disease,
* Not having chronic medication use that affects periodontal tissues (cyclosporine A, Phenytoin),
* Not having taken antioxidant supplements in the last 6 months.

Exclusion Criteria:

* Presence of any congenital craniofacial deformity (cleft lip and palate or any other craniofacial syndrome or deformity),
* Patients who have previously started or completed orthodontic treatment,
* Patients who have received periodontal treatment in the last 6 months,
* Acute illness,
* Systemic illness, mental illness, immunosuppressive medications, or immunodeficiency.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients coming to the Periodontology Clinic of Recep Tayyip Erdoğan University Faculty of Dentistry for routine periodontal treatment
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
Gingival crevicular fluid collection | Day 1
  After isolating the teeth with a cotton roll, supragingival plaque will be removed and a gentle airflow will be used to dry the teeth. GCF samples will be collected by inserting PerioPaper strips into the mesiobuccal gingival sulcus to a depth of approximately 1 mm for 30 seconds. A calibrated Periotron 8000 instrument will then be used to measure the total GCF volume. PerioPaper strips will then be stored at -80°C for future measurements.
Clinical Periodontal Parameters (Plaque Index) | Day 1
  Plaque Index (PI) This index is used to evaluate the amount of dental plaque accumulation on tooth surfaces. Each tooth's four surfaces (buccal, lingual, mesial, distal) are examined using a probe or visually. Each surface is scored from 0 to 3. The average score is calculated for each tooth.
  The overall plaque index is obtained by averaging the scores from all examined teeth.
  Score Description 0 No plaque.
  1. No visible plaque, but a slight film of plaque is detected when a probe is run along the gingival margin.
  2. Visible plaque along the gingival margin, forming a continuous band.
  3. Abundant plaque covering the gingival area and extending toward the middle of the tooth surface, including the interproximal spaces.
Periodontal Clinical Parametres (Papillary Bleeding Index) | Day 1
  Papillary Bleeding Index (PBI) This index is used to assess bleeding of the interdental papilla-an early sign of periodontal disease-in order to evaluate the degree of gingival inflammation.
  A periodontal probe is gently inserted into each interdental papilla (the triangular-shaped gum tissue between teeth). The probe is placed approximately 1-2 mm into the papilla and directed upward. Bleeding occurring within 10-30 seconds is observed and scored based on severity.
  The scores from all papillae are totaled and divided by the number of examined sites to obtain the average PBI score.
  Score Description 0 No bleeding
  1. Single-point, slight bleeding
  2. Thin line of blood
  3. Obvious and rapid bleeding across the entire papilla, slight spreading
  4. Severe, profuse bleeding that overflows the papilla, usually with evident inflammation
Periodontal Clinical Parametres (Bleeding on Probing Index) | Day 1
  Bleeding on Probing (BOP) Index This index is used to assess the presence and severity of gingival inflammation by observing bleeding after gentle pressure is applied to the gingival sulcus using a periodontal probe. A thin periodontal probe is gently inserted into the gingival sulcus with light pressure (approximately 20-25 grams). Bleeding occurring within 10-30 seconds is observed. Each measurement site is recorded as either "bleeding present" or "bleeding absent." Presence of bleeding is an early and sensitive indicator of gingival inflammation.
  Score Description 0 No bleeding
  1 Bleeding present (mild or severe)
Periodontal Clinical Parametres (Probing Pocket Depth) | Day 1
  Probing Pocket Depth (PPD)
  Using a Williams periodontal probe, the distance between the marginal gingival margin and the base of the periodontal pocket is measured in millimeters at six sites per tooth:
  mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual.
  All teeth are measured. The values obtained from each site are summed and then divided by the total number of sites measured.
  This gives the average probing depth for the individual.
  Measurement Interpretation 1-3 mm Healthy sulcus 4-5 mm Shallow to moderate pocket
  ≥6 mm Deep periodontal pocket (advanced disease)
Periodontal Clinical Parametres (Clinical Attachment Loss) | Day 1
  Clinical Attachment Loss (CAL)
  Using a Williams periodontal probe, the distance between the enamel-cementum junction and the base of the periodontal pocket is measured in millimeters at six sites per tooth:
  mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual.
  All teeth are measured. The values obtained from each site are summed and then divided by the total number of sites measured.
  This gives the average probing depth for the individual.
  CAL Value Interpretation 0-1 mm Healthy / minimal loss 2-3 mm Mild attachment loss 4-5 mm Moderate attachment loss
  ≥6 mm Severe attachment loss

SECONDARY OUTCOMES:
Determination of RANKL, OPG, TAS and TAC by ELISA | 4th month
  Frozen paper strips will be thawed and diluted with 200 μL of phosphate-buffered saline (pH 7.4). The mixture will then be centrifuged at 13,000 g for 10 min at 4 °C. RANKL, Osteoprotegerin (OPG), Total Oxidative Status (TOS), and Total Antioxidant Capacity (TAC) kits will be analyzed by ELISA. Results will be expressed as pg/μL.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology of the Faculty of Dentistry of Recep Tayyip Erdogan University, Rize, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No